CLINICAL TRIAL: NCT03262038
Title: A Randomized Double Blinded, Placebo-controlled Trial of IV Ondansetron to Prevent Pruritus in Children Who Receive Intrathecal Morphine
Brief Title: Does IV Ondansetron Prevent Pruritus After Intrathecal Morphine in Pediatric Patients?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed no difference between groups
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elizabeth Putnam, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HUM00124202
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-08

CONDITIONS: Pruritus; Nausea/Vomiting
Keywords: intrathecal morphine
MeSH Terms: conditions — Pruritus; Nausea; Vomiting | interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, placebo-controlled trial of ondansetron to prevent pruritus in children who receive intrathecal morphine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug (ondansetron/placebo) will be masked for all but the pharmacist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ondansetron IV (Experimental): Ondansetron IV X1 intraoperatively (0.1 mg/kg in 5 mLs) Ondansetron IV X 4 (Q 6 hrs for 24 hrs) (0.1 mg/kg in 5 mLs)
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Placebo Comparator: This arm will receive (in a blinded fashion) a volume-matched placebo intraoperatively X1 as well as IV every 6 hrs for 24 hours postoperatively. (X4)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Ondansetron — This arm will receive (in a blinded fashion) 0.1 mg/kg of Ondansetron IV made up to 5 mLs intra-operatively and Ondansetron IV 0.1 mg/kg made up to 5 mLs every 6 hours for 24 hours postoperatively.
  Arms: Ondansetron IV
Drug: Placebo Comparator — This arm will receive (in a blinded fashion) a volume-matched placebo intraoperatively as well as IV every 6 hrs for 24 hours postoperatively.
  Arms: Placebo

SUMMARY:
This is a prospective randomized, double-blind, placebo-controlled study to compare the incidence and intensity of ITM-induced pruritus and nausea/vomiting using pre-emptive IV ondansetron, followed by scheduled Around The Clock (ATC) ondansetron vs. our control group, where pruritus and PONV are treated with PRN only medications.

DETAILED DESCRIPTION:
Pruritus is one of the most common and bothersome side effects of intrathecal morphine (ITM) in children, with a reported incidence of 30-60%. Clinicians, who have witnessed unbearable itching and scratching in their young patients after intrathecal morphine, may be reluctant to offer this effective pain control to future patients, for fear of these unpleasant sequelae. A study previously found a 40% incidence of pruritus in young children who received intrathecal morphine for major urologic surgery.

This is a prospective randomized, double-blind, placebo-controlled study to compare the incidence and intensity of ITM-induced pruritus and nausea/vomiting using pre-emptive IV ondansetron, followed by scheduled Around The Clock (ATC) ondansetron vs. control group, where pruritus and PONV are treated with PRN only medications.

Enrollment of 3-17 year olds who are undergoing urologic or orthopedic operative procedures who are scheduled to receive low dose (4-5 mcg/kg) intrathecal morphine for pain management.

ELIGIBILITY:
Inclusion Criteria:

* 3-17 years
* weight </= 100kg
* scheduled for urologic or orthopedic procedure necessitating intrathecal morphine
* ability to use verbal or pictorial pain assessment tools and techniques
* informed consent and (if applicable) assent

Exclusion Criteria:

* Inability to use verbal or pictorial pain scoring scales
* hypersensitivity to selective 5-HT receptor antagonists
* diagnosed congenital long QT syndrome
* severe hepatic impairment
* pregnancy or nursing mothers

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Putnam, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ondansetron IV | Placebo
Started | 18 | 28
Completed | 18 | 27
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron IV | Placebo | Total
Number analyzed (Participants) | 18 | 27 | 45
Age, Customized [Mean (Full Range); unit: years] — mean [range]
  years | 8.3 [3.5 to 17.1] | 8.2 [3.7 to 16.7] | 8.3 [3.5 to 17.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 6 | 10 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Full Range); unit: kg] | 30.4 [16.4 to 64.8] | 34.0 [14.5 to 91.4] | 32.5 [14.5 to 91.4]
ASA 1, 2 [Count of Participants; unit: Participants] — Assesses physical status of a patient at the time of surgery. ASA 1: normal, healthy ASA 2: mild systemic disease (eg. asthma)
  Participants | 15 | 27 | 42
Surgical Service [Count of Participants; unit: Participants]
  Urology | 14 | 22 | 36
  Orthopedics | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pruritus
Description: number of participants with any incidence of pruritus
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron IV | Placebo
Number analyzed (Participants) | 18 | 27
Participants | 14 | 24
Statistical Analysis 1: Comparison: Ondansetron IV vs Placebo; Test type: Superiority; p = .412, Chi-squared

2. Primary Outcome: Severity of Pruritus
Description: number of participants who indicated mild pruritus (no treatment needed) or severe pruritus (treatment needed)
Time Frame: 24 hours
Population: Excludes those without any itch
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron IV | Placebo
Number analyzed (Participants) | 14 | 24
Participants
  Mild / no treatment needed | 1 | 4
  Severe / requiring treatment | 13 | 20
Statistical Analysis 1: Comparison: Ondansetron IV vs Placebo; Test type: Superiority; p = .633, Chi-squared

3. Secondary Outcome: Incidence of Post Operative Nausea or Vomiting
Description: number of participants with any incidence of postoperative nausea or vomiting
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron IV | Placebo
Number analyzed (Participants) | 18 | 27
Participants | 8 | 23
Statistical Analysis 1: Comparison: Ondansetron IV vs Placebo; Test type: Superiority; p = .007, Chi-squared

4. Secondary Outcome: Severity of Post Operative Nausea or Vomiting
Description: number of participants who Indicated mild post operative nausea or vomiting (no treatment needed) or severe postoperative nausea or vomiting(treatment needed)
Time Frame: 24 hours
Population: excludes those without any nausea vomiting
Measure: Count of Participants; unit: Participants
Arm/Group | Ondansetron IV | Placebo
Number analyzed (Participants) | 8 | 23
Participants
  Mild / no treatment required | 2 | 4
  Severe / requiring treatment | 6 | 19
Statistical Analysis 1: Comparison: Ondansetron IV vs Placebo; Test type: Superiority; p = .634, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were tracked through hospital discharge (approximately 24 hours)
Description: The AE reporting plan includes adverse events other than the two outcomes studied (AEs other than itch, nausea, or vomiting).
Arm/Group | Ondansetron IV | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/27
Other Adverse Events (participants affected / at risk) | 0/18 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03262038/Prot_SAP_001.pdf